CLINICAL TRIAL: NCT04611971
Title: A Phase 1, Single Center, Randomized, Controlled Platform Study Validating the Use of Candin As a Challenge Agent in Healthy Volunteers or Patients Given Concomitant Approved Interventions
Brief Title: A Study Validating the Use of Candin as a Challenge Agent in Healthy Participants - Intervention Specific Appendix 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR108910; 2020-002481-14 (EudraCT Number); NOPRODPANAP1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-10-29; First posted 2020-11-02 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Arm: Benlysta + Candin (Active Comparator): Participants will receive a single dose of Candin injection intradermally along with a saline solution of 0.9% sodium chloride (NaCl), and a single dose of Benlysta injection subcutaneously.
  Interventions: Drug: Benlysta; Drug: Candin
- Control Arm: Candin (No Intervention): All participants will receive a single dose of Candin injection intradermally along with a single dose of saline solution of 0.9% NaCl administered intradermally and no Benlysta.

INTERVENTIONS:
Drug: Benlysta — Benlysta injection will be administered subcutaneously.
  Other Names: Belimumab
  Arms: Active Arm: Benlysta + Candin
Drug: Candin — Candin will be administered intradermally along with NaCl solution.
  Arms: Active Arm: Benlysta + Candin

SUMMARY:
The purpose of this study is to characterize the delayed-type hypersensitivity (DTH) response at the site of Candin intradermal injection in the presence of a targeted immune pathway inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2, inclusive (BMI = weight/height^2), and body weight of no less than 50 kilograms (kg)
* Healthy on the basis of physical examination, medical history, and vital signs performed at screening. Any abnormalities, must be considered not clinically significant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Must be a non-smoker (not smoked for at least 6 months prior to screening) and has not used nicotine-containing products (example, nicotine patch) for 3 months prior to screening
* Has a negative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) coronavirus disease 2019 (COVID-19) reverse transcription polymerase chain reaction (RT-PCR) test within 72 hours prior to administration of study intervention
* A woman must be: a) not of childbearing potential; or b) of childbearing potential and practicing a highly effective method of contraception (failure rate of less than [<] 1 percent [%] per year when used consistently and correctly) and agrees to remain on a highly effective method while receiving study intervention and until 4 months after study intervention administration - the end of relevant systemic exposure. The investigator should evaluate the potential for contraceptive method failure (example, noncompliance, recently initiated) in relationship to the study intervention administration

Exclusion Criteria:

* History of liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic, or mucocutaneous disturbances
* Known allergies, hypersensitivity, or intolerance to Candin or its excipients
* Has an active, acute or chronic infection
* has a history of psychiatric disorders (depression, suicidal ideation and/or behavior including suicides)
* Has had prior exposure to belimumab or other B-cell activating factor (BAFF) inhibitors, such as tabalumab, atacicept, and telitacicept

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Presence and Size of Induration in Active Versus Control at the Candin Injection Site Compared to the Intra-individual Saline Control Injection Site Approximately 48 Hours After Candin Challenge | Day 8
  Number of participants with presence and size of induration in active versus control at the Candin injection site compared to the intra-individual saline control injection site approximately 48 hours after Candin challenge will be reported.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) in the Active Arm Versus the Control Arm | Up to 2 months
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Treatment-Emergent Serious Adverse Events (SAEs) in the Active Arm Versus the Control Arm | Up to 2 months
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants with TEAEs by Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC) with a Frequency Threshold of 5 Percent (%) or More in the Active Arm Versus the Control Arm | Up to 2 months
  Number of participants with TEAEs by MedDRA SOC with a frequency threshold of 5% or more in the active arm versus the control arm will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency